CLINICAL TRIAL: NCT04097769
Title: A Phase I, First-in-Human Study Evaluating the Safety, Tolerability, and Initial Efficacy of HX009 in Patients With Advanced Malignancies
Brief Title: The Safety, Tolerability, and Initial Efficacy of HX009 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Waterstone Hanxbio Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX009-I-01
Record Dates: First submitted 2019-08-28; First posted 2019-09-20 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: HX009
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX009 (Other): Study treatment: HX009 administered every 2 weeks (14 [±1] days) via intravenous infusion.
  Interventions: Drug: HX009

INTERVENTIONS:
Drug: HX009 — During study treatment, subjects will receive HX009 treatment via IV infusion once every 2 weeks at doses of 0.1, 0.3, 1, 2, 3, 5, and 7.5 mg/kg.
  Other Names: anti-PD-1/CD47 infusion protein

SUMMARY:
This is a first-in-human, multicenter, open-label, multiple-dose Phase I study to investigate the safety, tolerability, and initial efficacy of HX009 in subjects with advanced malignant tumors. The study will consist of a dose-escalation and dose-finding component to establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) and to evaluate the preliminary antitumor activity of HX009.

DETAILED DESCRIPTION:
The study will follow a 3+3 dose-escalation scheme enrolling cohorts of at least 3 subjects sequentially at escalating doses. During study treatment, subjects will receive HX009 treatment via intravenous infusion once every 2 weeks. Dose escalation will continue until identification of an MTD or the maximum dose is reached. Dose-limiting toxicities (DLTs) will be assessed from the first dose of study treatment (Day 1) until 28 days later (Day 29).

The study is divided into a screening period (28 days before first dose), treatment period (up to 24 months), and survival follow-up period. Safety will be evaluated throughout the study up until 90 (±7) days after the last dose of study treatment. Blood samples will be collected at regular intervals for pharmacokinetics (PK) and immunogenicity evaluation. Tumor evaluation (assessed by the Investigator in accordance with Response Evaluation Criteria in Solid Tumors Version 1.1 [RECIST 1.1] and immune RECIST [iRECIST]) to assess efficacy will start from the first dose and occur every 8 weeks in the first 12 months and every 12 weeks in the second 12 months and during the survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 18 to 70 years, inclusive.
2. Eastern Cooperative Oncology Group performance status of 0 to 1.
3. Histologically confirmed advanced malignant tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject refuses standard therapy.
4. At least 1 measurable tumor according to RECIST v1.1 (see Appendix 7 of the protocol).
5. Life expectancy ≥12 weeks.
6. A subject with a history of brain/meninges metastases who has received prior topical treatment (surgery/radiotherapy) before the start of the study and is clinically stable for at least 3 months is allowed (prior treatment with corticosteroids is permitted; however, if a subject requires systemic concomitant treatment with corticosteroids, they must be excluded).
7. Adequate organ function, as indicated by the following laboratory values, within 14 days before signing informed consent:

   Hematology
   * Hemoglobin ≥100 g/L (no blood transfusion is allowed within 14 days before signing informed consent)
   * Absolute neutrophil count ≥1.5 × 109/L
   * Platelet count ≥100 × 109/L Biochemistry
   * Total bilirubin ≤1.5 × upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN (ALT and AST ≤5 × ULN for subjects with liver metastases)
   * Serum creatinine ≤1 × ULN
   * Prothrombin time/international normalized ratio ≤1.5 × ULN or activated partial thromboplastin time ≤1.5 × ULN (for subjects on anticoagulants, prothrombin time or activated partial thromboplastin time must be within the normal range for anticoagulants).
8. Male subject: must agree to use contraception as detailed in Appendix 5 of this protocol during the treatment period and for at least 12 months after the last dose of the study treatment.

   Female subject: must not be pregnant; or must not be of childbearing potential as defined in in Appendix 5; or if of childbearing potential, must agree to use highly effective birth control methods during the study treatment period and for at least 12 months after the last dose of the study treatment.
9. Voluntarily agrees to participate by giving written informed consent and is willing and able to comply with protocol and scheduled visits.

Exclusion Criteria:

1. For subjects who have received prior anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4):

   * Subjects must not have received anti-PD-1, anti-PD-L1, anti-CTLA-4, CD47, or any other immunotherapy or immune-oncology agent within 4 weeks of the first dose study treatment
   * Subjects must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy
   * Any adverse events reported while receiving prior immunotherapy must have completely resolved or resolved to Grade 1 prior to screening for this study.
2. Prior malignancy active within the previous 2 years except for the tumor for which a subject is enrolled in the study and locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
3. Allergic to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components.
4. Receipt of any immunotherapy, or investigational anticancer therapy within 4 weeks prior to the first dose of study treatment; in the case of mAbs (for investigational use or immunotherapy), 6 weeks prior to the first dose of study treatment.
5. Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy (except for subjects with metastatic prostate cancer on androgen deprivation treatment eg, goserelin, leuprorelin) for cancer. Concurrent use of hormones for noncancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable. NOTE: Local treatment of isolated lesions for palliative intent is acceptable (eg, by local surgery or local radiotherapy).
6. Radiation therapy (localized radiation therapy for therapeutic purpose is allowed) within 4 weeks of the first dose of study treatment.
7. Female subject who is pregnant or lactating.
8. Tests positive for human immunodeficiency virus, or has active hepatitis B virus or hepatitis C virus.
9. Active, or history of, autoimmune disease (within the past 2 years) that may recur (eg, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, etc) or are at high risk (eg, receiving an immunosuppressive treatment for an organ transplant); however, subjects with the following are allowed to enroll:

   * Type I diabetes that is stable after a fixed dose of insulin
   * Only requiring hormone replacement therapy for autoimmune hypothyroidism
   * Skin disease that does not require treatment such as eczema, rash that accounts for <10% of the body surface, psoriasis without ophthalmic symptoms.
10. Planning major surgery during the study including the screening period.
11. Requiring systemic corticosteroids (dose equivalent to >10 mg prednisone/day) or other immunosuppressive drugs within 14 days before the first dose of study treatment or during the study. The following are allowed:

    * Use of topical or inhaled glucocorticoids
    * A brief course of corticosteroids (≤7 days) for prophylaxis or for treatment of non autoimmune conditions.
12. Active peptic ulcer, incomplete intestinal obstruction, active gastrointestinal bleeding, and perforation.
13. Lung disease, interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease, interstitial pneumonia, etc.
14. Uncontrolled stable systemic diseases such as cardiovascular and cerebrovascular diseases, diabetes, high blood pressure, etc.
15. History of infection with human immunodeficiency virus, or other acquired, congenital immunodeficiency disease, or history of organ transplantation, or history of stem cell transplantation.
16. Current, or history of, tuberculosis or evidence of latent tuberculosis infection: positive QuantiFERON-TB Gold assessment at screening.
17. Severe infections within 4 weeks before the first dose of study treatment, or active infections within 2 weeks before the first dose that require oral or intravenous antibiotics.
18. Cancerous meningitis.
19. Has received hematopoietic stimulating factors such as colony stimulating factor and erythropoietin within 2 weeks before the first dose of study treatment.
20. Use of any live vaccines within 4 weeks before the first dose of study treatment.
21. Any major surgery within 4 weeks before the first dose of study treatment (except for diagnostic surgery).
22. A history of psychotropic substance abuse who is unable to quit or who has a history of mental disorders.
23. Other severe, acute or chronic medical or psychiatric diseases or laboratory abnormalities that, in the Investigator's opinion, may increase the study-related risks or interfere with the interpretation of the findings.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | All AEs up to 90 days after the last dose of study drug
  An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product.
Number of Participants With Dose-Limiting Toxicities (DLT) of HX009 | At the end of Cycle2(each cycle is 14 days)
  Severity of adverse events (AEs) was graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. For the purpose of dose escalation, any of the following AEs occurring during the DLT observation period that were attributable to one or both study drugs were classified as DLTs.

SECONDARY OUTCOMES:
Time for Cmax (Tmax) of HX009 | Approximately 2 years
  Time to reach HX009 maximum observed serum concentration.
Terminal Half-life （t½）of HX009 | Approximately 2 years
  HX009 terminal half-life.
Area Under the Serum Concentration-time Curve (AUC) | Approximately 2 years
  HX009 area under the serum concentration-time curve .
Number of Participants With Positive Anti-Drug Antibody (ADA) of HX009 | Cycles 1, 2, 3, 4, 5, 6, 7, 9, 13, and 17, and then every 8 cycles, Day 1: within 60 minutes before the start of the infusion(each cycle is 14 days)
  ADA blood samples were assayed for anti-HX009 antibodies.
Objective response rate(ORR) Per Investigator Assessment Using RECIST 1.1 | Approximately 2 years
  The ORR, using RECIST 1.1 criteria, was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) at any time during the study, based on Investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul de Souza, Principal Investigator — St George Private Hospital
Locations (1):
- St George Private Hospital, Kogarah, New South Wales, Australia